CLINICAL TRIAL: NCT06654973
Title: The Singapore Platform for Controlled Human Infections With SARS-CoV-2
Brief Title: Singapore SARS-CoV-2 Human Challenge Study
Acronym: Sing-CoV
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: A*Star (Other); Duke-NUS Graduate Medical School (Other)
Responsible Party: Principal Investigator, Barnaby Young, Head of Singapore Infectious Disease Clinical Research Network, Tan Tock Seng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023/00911
Record Dates: First submitted 2024-10-09; First posted 2024-10-23 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: COVID 19
Keywords: SARS-CoV-2; Human challenge study; Delta variant; Correlates of protection; Determinants of breakthrough infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SARS-CoV-2 Delta human infection challenge (Experimental): GMP-produced Delta SARS-CoV-2 virus will be given to participants via intranasal drops.
  Interventions: Other: GMP-produced SARS-CoV-2 Delta strain

INTERVENTIONS:
Other: GMP-produced SARS-CoV-2 Delta strain — The challenge virus used in Sing-CoV study is the same as that used in COVHIC002 study. It was originally obtained in mid 2021 from a nose-throat swab from an otherwise healthy young adult with mild COVID-19 in the community. The procedure for isolation, storage, preparation, and administration of challenge virus in this study (Sing-CoV and COVHIC002) is the same as used in the first SARS-CoV-2 human challenge study (COVHIC001) at Imperial College London and the same as used in the COV-CHIM01 (NCT04864548) SARS-CoV-2 human challenge study at University of Oxford.

SUMMARY:
The goal of this study is to conduct a safe SARS-CoV-2 Delta variant human infection challenge in adult healthy volunteers. The main objectives are to:

* Induce laboratory confirmed infection in up to 70% of participants
* Confirm the safety profile as measured by the occurrence of adverse events (AEs) and serious adverse events (SAEs) from the day of viral challenge (Day 0) up to Day 28 follow-up.

Participants will be given the GMP-produced Delta SARS-CoV-2 virus via intranasal drops using the optimized conditions established in the "Development of a SARS-CoV-2 Delta variant human infection challenge model" (COVHIC002) Human Challenge Study being conducted in the UK. A safe and well-tolerated human challenge model with the SARS-CoV-2 Delta variant will be established in Singapore. This model will be used to accelerate next-generation vaccine development and to determine the factors associated with altered clinical and virological outcomes; correlates of protection; and targets for the development of novel vaccines, therapeutics, and diagnostics.

DETAILED DESCRIPTION:
Human challenge studies involve the deliberate infection of volunteers to allow detailed investigation of host-pathogen interactions and the effect of interventions. The strength of these studies lies in their highly controlled nature. Carefully selected participant groups are inoculated with standardised amounts of a well-characterised virus. This enables exact longitudinal measurement of viral kinetics, immunological responses, transmission dynamics and the duration of infectious shedding. By giving all study participants the same virus at the same dose and under the same conditions, confounding by virus strain, dose, and exposure is controlled. Host factors associated with inter-individual differences in clinical outcome as well as the effect of interventions can then be robustly inferred.

The Human Challenge study contrasts with even the most well-controlled field trials, including household contact studies. In natural infection, the virus quasi-species (i.e., mixture of slightly differing virus particles), dose, timing and conditions of exposure cannot be known, and contacts are only identified following diagnosis of the index case. At this time, secondary exposure has almost always already occurred, thus missing transmission events as well as the early phase of infection. Human challenge is therefore the only study design where the earliest pre-symptomatic changes post infection may be studied. These early time-points are critical to understanding how some people who are exposed to a virus resist infection and to delineate early infectiousness and transmissibility.

The first SARS-CoV-2 human challenge study (COVHIC001) was conducted in 2021 and showed no serious safety concerns after inoculating 36 healthy, unvaccinated, young adults with a pre-Alpha "Wuhan" strain of SARS-CoV-2. A follow up human challenge study with a Delta variant (COVHIC002) is currently ongoing in the UK. COVHIC002 will determine and optimise the conditions for a safe human challenge model with the SARS-CoV-2 Delta variant. These conditions will subsequently be applied in this companion study, Sing-CoV.

Importantly, a model of vaccine breakthrough infection will have a substantially improved safety profile compared with the first (seronegative) study as:

1. The risk of severe disease and protracted symptoms among healthy volunteers are substantially reduced by vaccination;
2. Highly effective anti-virals are available as rescue therapy;
3. Data from the SARS-CoV-2 human challenge studies (both COVHIC001 and COVHIC002) underpin the design of the Sing-CoV study and supports robust informed consent.

Recent SARS-CoV-2 variants-of-concern (VOC; Delta and Omicron) have shown high rates of vaccine breakthrough infection, indicating that human challenge with these strains may be optimised as a platform for the rapid testing of vaccines and therapeutics in small numbers of participants despite pre-existing immunity, especially between waves of the pandemic, when occurrence of natural disease is relatively uncommon. This will enable efficient early-stage testing of the many vaccine and antiviral candidates in development so that the most promising can go forward quickly enough to large-scale field efficacy trials to meaningfully tackle the ongoing pandemic.

Thus, in the short term, a Delta human challenge model will uniquely enable:

1. A model of breakthrough infection that can be used to assess transmission blocking potential of new vaccines and treatments.
2. Identification of the immune factors associated with susceptibility to breakthrough infection.
3. Studies that can uniquely provide proof-of-principle efficacy data for vaccine candidates that confer cross-strain protection.

Establishing the capability to perform SARS-CoV-2 human challenge studies in Singapore will be highly significant. Firstly, this will facilitate development of therapeutics and vaccines in the region; secondly, it will ensure inferences drawn from SARS-CoV-2 human challenge studies are applicable to people of Asian ethnicity; and thirdly, it will support capacity development in the region where future coronavirus pandemics (like SARS-CoV-1 and SARS-CoV-2) are expected to originate.

ELIGIBILITY:
Inclusion Criteria:

1. An informed consent form (ICF) has been signed and dated by the participant, an investigator, and a witness
2. Adults age between 21 and 30 years inclusive (at the time of consent)
3. Evidence of having had a complete primary COVID-19 vaccination course as recommended by the Ministry of Health*, with the last vaccination at least 14 days before enrolment
4. Sero-suitable based on the pre-screening serology result 5a) Female participants must be willing and able to use contraception from 2 weeks before the scheduled date of viral challenge until 6 months after receipt of the final dose of study virus. Negative urine pregnancy tests will be required at screening, and on admission to the quarantine unit a negative serum beta human chorionic gonadotropin (β-hCG) is required prior to inoculation.

5b) Male participants who are willing to use one of the contraception methods described in the study protocol, from the time of the date of viral challenge, for 6 months.

6) In good health with no history of clinically significant medical conditions (as described in Exclusion criteria) that would interfere with subject safety, as defined by medical history, physical examination and routine laboratory tests, ECG, and Chest X-Ray and determined by the Investigator at an admission evaluation.

7) Willing and able to commit to participation in the study.

Exclusion Criteria:

1. History or evidence of any clinically significant or currently active cardiovascular, (including thromboembolic events), respiratory, dermatological, gastrointestinal, endocrine, haematological, hepatic, immunological, rheumatological, metabolic, urological, renal, neurological, psychiatric illness. Specifically:

   1. Participants with any history of physician diagnosed and/or objective test confirmed asthma, chronic obstructive pulmonary disease, pulmonary hypertension, reactive airway disease, or chronic lung condition of any aetiology or who have experienced:

      * Significant/severe wheeze in the past
      * Respiratory symptoms including wheeze which has ever resulted in hospitalisation
      * Known bronchial hyperreactivity to viruses
   2. History of thromboembolic, cardiovascular or cerebrovascular disease
   3. History or evidence of diabetes mellitus
   4. Any concurrent serious illness including history of malignancy that could interfere with the aims of the study or a participant completing the study. Basal cell carcinoma within 5 years of treatment or with evidence of recurrence is also an exclusion
   5. Migraine with associated neurological symptoms such as hemiplegia or vision loss. Cluster headache/migraine or prophylactic treatment for migraine
   6. History or evidence of autoimmune disease or known immunodeficiency of any cause.
   7. Other major disease that, in the opinion of the Investigator, could interfere with a participant completing the study and necessary investigations.
2. Any significant abnormality altering the anatomy or function of the nose or nasopharynx in a substantial way (including loss of or alterations in smell or taste), a clinically significant history of epistaxis (large nosebleeds) within the last 3 months, nasal or sinus surgery within 6 months of inoculation.
3. Clinically active rhinitis (including hay fever) or history of moderate to severe rhinitis, or history of seasonal allergic rhinitis likely to be active at the time of inclusion into the study and/or requiring regular nasal corticosteroids on an at least weekly basis, within 30 days of admission to quarantine.
4. History of anaphylaxis and/or a history of severe allergic reaction or significant intolerance to any food or drug, as assessed by the PI.
5. Significant history or presence of drug or alcohol misuse
6. Current use of any drugs taken through the nasal or inhaled route
7. Psychiatric illness including participants with a history of depression and/or anxiety with associated severe psychiatric comorbidities, for example psychosis.

   Consider exclusion in the following cases: (a) Participants with history of anxiety-related symptoms of any severity within the last 2 years if the Generalized Anxiety Disorder-7 score is ≥4; (b)Participants with a history of depression of any severity within the last 2 years if the Patient Health Questionnaire-9 score is ≥4. (c) severe claustrophobia
8. Current active smokers: equivalent to >5 cigarettes per week, including use of tobacco in any form (e.g., smoking or chewing) or other nicotine-containing products in any form (e.g., gum, patch) or electronic cigarettes.

   Ex-smokers: Participants who have smoked >5 pack years at any time [5 pack years is equivalent to one pack of 20 cigarettes a day for 5 years]. Ex-smokers that have smoked <5 pack years at any time must not have smoked in the last 3 months.
9. Family history of 1st degree relative aged 50 years or less with sudden cardiac or unexplained death
10. Personal or Family History of unexpectedly severe COVID-19 (including a personal history of COVID-19 pneumonia), severe adverse response to any other viral disease e.g., Guillain-Barré, or a family history (described as a 1st degree relative) with clotting disorders
11. A total body weight of ≤ 45kg and a Body Mass Index (BMI) ≤18 kg/m2 and ≥28 kg/m2. The upper limit of BMI may be increased to 30kg/m2 at the PI's discretion, in the case of physically fit muscular individual
12. Venous access deemed inadequate for the phlebotomy demands of the study.
13. Any clinically significant abnormal finding on screening biochemistry, haematology and microbiology blood tests or urinalysis apart from minor deviations which are clinically acceptable and approved by the investigator.

    Any of the following:
    * Elevated HbA1C
    * Positive HIV, active/chronic hepatitis B or C test.
14. A forced expiratory volume in 1 second (FEV1) and a forced vital capacity (FVC) <80% of predicted value calculated using ATS/ERS guidance
15. Twelve-lead ECG recording with clinically relevant abnormalities as judged by the study investigator.
16. History of, or currently active symptoms suggestive of upper or lower respiratory tract infection (including reduced sense of taste and smell, raised body temperature and/or persistent cough) within 4 weeks prior to viral challenge.
17. Presence of cold-like symptoms and/or fever (defined as participant presenting with a temperature reading of >37.9ºC) on Day -1 and/or pre-challenge on Day 0.
18. Evidence of any respiratory virus infection (on Respiratory PCR from upper respiratory tract sample) on admission to the quarantine unit, prior to challenge virus inoculation.
19. Receipt of a live vaccine within 60 days prior to the planned date of viral challenge, a non-live vaccine within 30 days prior to the planned date of viral challenge or intention to receive any vaccination(s) before the day 28 follow-up visit.
20. Receipt of blood or blood products, or loss (including blood donations) of 550 mL or more of blood during the 3 months prior to the planned date of viral challenge or planned during the 3 months after the final visit.
21. Medications:

    1. Use of any medication or product (prescription or over the counter), for symptoms of allergic rhinitis, nasal congestion or respiratory tract infections or dermatitis/eczema including the use of regular nasal or medium-high potency dermal corticosteroids, and antibiotics within 7 days prior to the planned date of viral challenge apart from those described in Table 7, Permitted Medication or agreed by the investigator
    2. Receipt of any investigational drug within 3 months prior to the planned date of viral challenge
    3. Receipt of systemic (intravenous and/or oral) glucocorticoids or systemic antiviral drugs within 6 months prior to the planned date of viral challenge.
    4. Over the counter medications (e.g., paracetamol or ibuprofen) where the dose taken over the preceding 7 days prior to the planned date of viral challenge had exceeded the maximum permissible 24-hour dose (e.g., >4g per day of paracetamol over the preceding week).
    5. Chronically used medications, including any medication known to be a moderate/potent inducer or inhibitor of cytochrome P450 enzymes, within 21 days prior to the planned date of viral challenge.
    6. Participants who have received any systemic chemotherapy agent, immunoglobulins, or other cytotoxic or immunosuppressive drugs at any time.
22. Previous participation in a SARS-CoV-2 vaccine trial of a currently unapproved/unlicensed vaccine in Singapore
23. Participant is mentally or legally incapacitated in the opinion of the Investigator.
24. Females who:

    1. Are breastfeeding within 6 months of study commencement, or
    2. Had been pregnant within 6 months prior to the study, or
    3. Had a positive pregnancy test at any point during screening or prior to inoculation with challenge virus
25. Anyone who is first degree related to anyone who is a delegated member of the research team.
26. Any other reason that the Investigator considered made the participant unsuitable to participate.
27. Participants with no knowledge of their family history.

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2025-12-29 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To identify a safe dose of SARS-CoV-2 in healthy volunteers in Singapore, suitable for future intervention studies | From day of viral challenge (Day 0) to Day 28 follow-up visit
  To evaluate the safety of a SARS-CoV-2 challenge in healthy participants by assessing:
  * Occurrence of unsolicited AEs post-viral challenge (Day 0) up to the Day 28 follow up visit.
  * Occurrence of SAEs related to the viral challenge from the viral challenge (Day 0) up to the Day 28 follow up visit.
To identify an infectious dose of SARS-CoV-2 in healthy volunteers in Singapore, suitable for future intervention studies | From day 2 post-inoculation to day of discharge from quarantine (Day 10 for uninfected participants or Day 14 for infected participants)
  To determine the attack rate of the Delta variant SARS-CoV-2 inoculum dose of TID 1x106 in sero-selected participants. Laboratory confirmed infection is defined as:
  • Two quantifiable greater than lower limit of quantification (≥LLOQ) RT-PCR measurements from mid turbinate and/or throat samples, reported on 2 or more consecutive timepoints, starting from Day 2 post-inoculation and up to discharge from quarantine.

SECONDARY OUTCOMES:
To further assess SARS-CoV-2 viral infection rates in upper respiratory samples in healthy volunteers | From day of viral challenge (Day 0) to day of discharge from quarantine (Day 10 for uninfected participants or Day 14 for infected participants)
  To assess the incidence of laboratory confirmed infection rates using a) mid turbinate samples, b) throat swabs, and c) both mid turbinate and throat swabs.
To assess the incidence of symptomatic SARS-CoV-2 infection, in healthy volunteers | From day of viral challenge (Day 0) to day of discharge from quarantine (Day 10 for uninfected participants or Day 14 for infected participants)
  To assess the incidence of lab-confirmed symptomatic SARSCoV-2 infection using a) mid turbinate samples, b) throat swabs, and c) both mid turbinate and throat swabs.
To assess the SARS-CoV-2 viral dynamics in upper respiratory samples in healthy volunteers | Day of inoculation (Day 0) to day of discharge from quarantine (Day 10 for uninfected participants or Day 14 for infected participants)
  To assess viral dynamics using a) mid turbinate samples, and b) throat swabs, as measured by qPCR.
To assess SARS-CoV-2 induced symptoms, in healthy volunteers | Day of inoculation (Day 0) to day of discharge from quarantine (Day 10 for uninfected participants or Day 14 for infected participants)
  Sum total symptoms diary card score: sum total clinical symptoms (TSS) as measured by graded symptom scoring system, starting one day post-viral challenge (Day 1) up to discharge from quarantine.
To assess the incidence of SARS-CoV-2 illness, in healthy volunteers | Day of inoculation (Day 0) to discharge from quarantine (Day 10 for uninfected participants or Day 14 for infected participants)
  The incidence of:
  * Upper Respiratory Tract illness (URTI)
  * Lower Respiratory Tract illness (LRTI)
  * Systemic illness (SI)
  * Febrile illness (FI)
  * Proportion of participants with Grade 3 symptoms on any occasion at any time from the last assessment on Day 0 to discharge from quarantine
  * Proportion of participants with Grade 2 or higher symptoms on any occasion at any time from the last assessment on Day 0 to discharge from quarantine
  * Proportion of participants with Grade 2 or higher Symptoms on two separate occasions at any time from the last assessment on Day 0 to discharge from quarantine
  * Proportion of participants with any symptom (grade >=1) on any occasion at any time from the last assessment on Day 0 to discharge from quarantine
  * Proportion of participants with any symptom (grade >=1) on two separate occasions at any time from the last assessment on Day 0 to discharge from quarantine

OTHER OUTCOMES:
To explore the changes in smell (anosmia/parosmia) through infection. | Day of inoculation (Day 0) to Day 28 follow up
  The University of Pennslvania Smell Identification Test (UPSIT) will be used. It is provided as booklets containing a series of cards that the participants scratch and smell then asked to identify the odours. The test provides an index of absolute dysfunction (ie, anosmia, severe microsmia, moderate microsmia, mild microsmia, normosmia, factitious), as well as relative dysfunction based upon age and gender-adjusted normative percentile ranks. The total number of odorant stimuli out of 40 that is correctly identified serves as the test measure. Scores on this test correlate well with other types of olfactory tests, including threshold tests. The UPSIT is designed to be self-administered after explanation of the test by study staff and will be performed once before virus inoculation and then approximately every third day starting from Day 1, though the test can be conducted more frequently at the discretion of the Investigator.
To explore the safety of a SARS-CoV-2 human challenge model in healthy adults | Day of inoculation (Day 0) to Day 28 follow up
  To explore safety related measures of SARS-CoV-2 challenge in healthy participants by assessing the occurrence of haematological and biochemical laboratory abnormalities during the quarantine period.
To explore the SARS-CoV-2 viral infection rates in saliva in healthy volunteers | From Day 2 post-inoculation to discharge from quarantine (Day 10 for uninfected participants or Day 14 for infected participants)
  To measure the laboratory confirmed infection rates, as defined by:
  * Occurrence of at least two quantifiable (≥LLOQ) qPCR measurements, reported on 2 or more consecutive time points, starting from Day 2 post-inoculation and up to discharge from quarantine.
  * Occurrence of at least two detectable (≥LLOD) qPCR measurements, reported on 2 or more consecutive time points, starting from Day 2 post-inoculation and up to discharge from quarantine.
  * Occurrence of at least one quantifiable (≥LLOQ) SARS-CoV-2 viral cell culture measurement, starting from Day 2 post-inoculation and up to discharge from quarantine.
To explore the SARS-CoV-2 viral dynamics in saliva in healthy volunteers | From Day 1 post-inoculation up to discharge from quarantine (Day 10 for uninfected participants or Day 14 for infected participants)
  To assess viral dynamics in saliva by qPCR.
To explore SARS-CoV-2 viral infection in stool of healthy volunteers | From Day 1 post-inoculation up to discharge from quarantine (Day 10 for uninfected participants or Day 14 for infected participants)
  To measure SARS-CoV-2 excretion in the stool by:
  • Virus detection and quantification using qRT-PCR
To explore the changes in humoral immunity after SARS-CoV-2 challenge | Up to Day 360 post-inoculation
  Assays performed on blood, stool and mucosal samples to assess humoral immunity / systems serology SARS-CoV-2 (for example: SARS-CoV-2 neutralizing titres, ELISAs to IgG, IgM, IgA, sIgA, ADCC)
To explore the proteomic changes after SARS-CoV-2 challenge | Up to Day 360 post-inoculation
  Assays performed on blood, stool and mucosal samples to assess proteomic levels and changes (for example, cytokine and chemokines).
To explore the changes in cellular immunity after SARS-CoV-2 challenge | Up to Day 360 post-inoculation
  Assays performed on blood, stool and mucosal samples include cellular cell quantification and quality of immunity (for example T and B cell frequencies, phenotypes, and functionality assays, ELISPOTs, ICS).
To explore the transcriptomic changes after SARS-CoV-2 challenge | Up to Day 360 post-inoculation
  Assays performed on blood, stool and mucosal samples to measure transcriptome levels and changes (for example, RNAseq, single cell RNAseq, microarray, PCR)
To explore environmental contamination in the SARS-CoV-2 human challenge model in healthy adults | Day of admission (Day -1) to day of discharge from quarantine (Day 10 for uninfected participants or Day 14 for infected participants)
  Air samples, exhaled breath samples with the use of a face mask or G-II exhaled breath collector, and surface swab samples will be used for virus detection and quantification.
To explore changes in the vasculature during SARS-CoV-2 infection in healthy adults | Up to Day 360 post-inoculation
  To measure changes in endothelial function during SARS-CoV-2 infection:
  • To assess levels of endothelial derived mediators (e.g., prostacyclin, endothelin-1, nitric oxide) in the plasma
To explore the performance of antigen rapid tests (ART) during SARS-CoV-2 infection of healthy adults | Day of admission (Day -1) to day of discharge from quarantine (Day 10 for uninfected participants or Day 14 for infected participants)
  To explore the performance of antigen rapid tests performed by participants themselves following manufacturer's instructions (no additional training) in comparison with SARS-CoV-2 PCR and culture

CONTACTS AND LOCATIONS:
Overall Officials: Barnaby E Young, MB BChir, PhD, Principal Investigator — National Centre for Infectious Diseases
Locations (1):
- National Centre for Infectious Diseases, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
All study findings and documents will be regarded as confidential. The investigators and other study personnel must not disclose such information without prior written approval from the PI. Participant confidentiality will be strictly maintained to the extent possible under the law and local hospital policy. Identifiable information will be removed from any published data.

REFERENCES:
- [Background] Zhou J, Singanayagam A, Goonawardane N, Moshe M, Sweeney FP, Sukhova K, Killingley B, Kalinova M, Mann AJ, Catchpole AP, Barer MR, Ferguson NM, Chiu C, Barclay WS. Viral emissions into the air and environment after SARS-CoV-2 human challenge: a phase 1, open label, first-in-human study. Lancet Microbe. 2023 Aug;4(8):e579-e590. doi: 10.1016/S2666-5247(23)00101-5. Epub 2023 Jun 9. PMID 37307844
- [Background] Killingley B, Mann AJ, Kalinova M, Boyers A, Goonawardane N, Zhou J, Lindsell K, Hare SS, Brown J, Frise R, Smith E, Hopkins C, Noulin N, Londt B, Wilkinson T, Harden S, McShane H, Baillet M, Gilbert A, Jacobs M, Charman C, Mande P, Nguyen-Van-Tam JS, Semple MG, Read RC, Ferguson NM, Openshaw PJ, Rapeport G, Barclay WS, Catchpole AP, Chiu C. Safety, tolerability and viral kinetics during SARS-CoV-2 human challenge in young adults. Nat Med. 2022 May;28(5):1031-1041. doi: 10.1038/s41591-022-01780-9. Epub 2022 Mar 31. PMID 35361992